CLINICAL TRIAL: NCT05018650
Title: A Prospective, Randomized, Controlled, Interventional Clinical Trial to Evaluate the Safety and Effectiveness of the Route 92 Medical MonoPoint® Reperfusion System for Aspiration Embolectomy in Acute Ischemic Stroke Patients (SUMMIT MAX)
Brief Title: A Randomized, Controlled Trial to Evaluate the Safety and Effectiveness of the Route 92 Medical Reperfusion System (SUMMIT MAX)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Route 92 Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP 0974
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Route 92 Medical Monopoint Reperfusion System (Experimental): Aspiration thrombectomy with the Route 92 Medical HiPoint 88 and HiPoint 70 Reperfusion Catheters as part of the Monopoint Reperfusion System to treat acute ischemic stroke
  Interventions: Device: Route 92 Medical Reperfusion System
- Aspiration Predicate (Active Comparator): Aspiration thrombectomy with a predicate aspiration device to treat acute ischemic stroke
  Interventions: Device: Route 92 Medical Reperfusion System

INTERVENTIONS:
Device: Route 92 Medical Reperfusion System — Mechanical thrombectomy for acute ischemic stroke patients with large vessel occlusions will be performed with direct aspiration consisting of navigating a large-bore catheter up to the face of the clot and initiating vacuum suction.

SUMMARY:
The SUMMIT MAX study is a prospective, randomized, controlled, interventional clinical trial to evaluate the safety and effectiveness of the Route 92 Medical MonoPoint® Reperfusion System with the Hi Point 88 and HiPoint 70 Reperfusion Catheters for aspiration thrombectomy in acute ischemic stroke patients.

DETAILED DESCRIPTION:
The purpose of the SUMMIT MAX study is to obtain the safety and effectiveness data necessary to demonstrate substantial equivalence of the Route 92 Medical Reperfusion System with a predicate aspiration device to support a 510(k) application to the U.S. Food and Drug Administration (FDA) under the classification product code, NRY.

ELIGIBILITY:
Inclusion Criteria:

1. The consent process has been completed and documented according to applicable country regulations and as approved by the IRB / Ethics Committee
2. Age >=18 years
3. Patient presenting with clinical signs consistent with an acute ischemic stroke
4. Baseline National Institutes of Health Stroke Scale (NIHSS) score >= 6
5. Pre-stroke modified Rankin Score (mRS) <= 2
6. Baseline ASPECTS >= 6
7. Endovascular treatment initiated (defined as time of groin puncture) within 8 hours from time last known well
8. If indicated, thrombolytic therapy shall be initiated per clinical guidelines. If eligible for thrombolytic therapy, subjects should be treated as soon as possible and lytic use should not be delayed regardless of potential eligibility for mechanical neurothrombectomy.
9. The patient is indicated for aspiration neurothrombectomy with the Route 92 Medical Reperfusion System as determined by the Investigator
10. Angiographic confirmation of a large vessel occlusion of the M1 segment of the middle cerebral artery or distal internal carotid artery

Exclusion Criteria:

1. Known pregnancy or breast feeding
2. In the Investigator's opinion, any known comorbidity (including COVID-19 positivity) that may complicate treatment or prevent improvement or follow-up
3. Known serious, advanced, or terminal illness with anticipated life expectancy < 12 months
4. Known history of severe allergy to contrast medium
5. Known to have suffered a stroke in the past 90 days
6. Known connective tissue disorder affecting the arteries (e.g. Marfan syndrome, Ehlers-Danlos syndrome)
7. Any known previous cerebral hemorrhagic event
8. Any known pre-existing coagulation deficiency
9. Known hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR >3.0
10. Known baseline platelet count <50,000/µL
11. Known baseline blood glucose of <50 mg/dL or >400 mg/dL
12. Known to be participating in another study involving an investigational device or drug
13. Clinical symptoms suggestive of bilateral stroke or stroke in multiple territories.
14. Computed Tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of recent/ fresh cerebral hemorrhage (the presence of microbleeds is allowed)
15. Baseline CT or MRI showing intracranial tumor (except small meningioma <= 2cm) or significant mass effect with midline shift due to the tumor
16. Presumed septic thrombus, or suspicion of bacterial endocarditis
17. Inability to access the cerebral vasculature in the opinion of the neurointerventional team
18. Unlikely to be available for a 90-day follow-up (e.g. no fixed home address)
19. Evidence of arterial dissection in a vessel that must be traversed
20. Evidence of high-grade stenosis or occlusion (i.e., tandem occlusion) in a vessel that must be traversed
21. Known active or recent history of cocaine or methamphetamine abuse (within last 6 months)
22. Known history or presence of aneurysm or arteriovenous malformation (AVM) in the territory of the target lesion
23. For all patients, severe sustained hypertension with SBP >200 and/or DBP >120; for patients treated with a lytic, sustained hypertension despite treatment with SBP >185 and/or DBP >110
24. Treatment with heparin within 48 hours with a partial thromboplastic time more than two times the laboratory normal or treatment with any LMWH within 48 hours
25. Renal failure with serum creatinine >3.0 or Glomerular Filtration Rate (GFR) <30
26. Ongoing seizure due to stroke
27. Evidence of active systemic infection
28. Known cancer with metastases
29. Angiographic evidence of a dissection in the extracranial or intracranial cerebral arteries
30. Arterial stenosis requiring balloon angioplasty or stenting at the time of the procedure
31. Angiographic evidence of multiple cerebrovascular occlusions (e.g., bilateral anterior circulation, anterior/posterior circulation, tandem occlusions)
32. Angiographic evidence of known or suspected underlying intracranial vasculopathy or atherosclerotic lesions responsible for the target occlusion
33. Angiographic evidence or suspicion of aortic dissection
34. Angiographic evidence of an aneurysm or arteriovenous malformation (AVM) in the territory of the target lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with successful arterial revascularization defined as a modified Thrombolysis in Cerebrovascular Infarction (mTICI) score of 2b or greater | During procedure
  mTICI of 2b or greater indicates successful reperfusion following blood clot removal
Incidence of all symptomatic intracerebral hemorrhage (sICH) | within 24 hours post-procedure
  Evaluation of sICH per von Kummer et al

CONTACTS AND LOCATIONS:
Overall Officials: Guilherme Dabus, MD, Principal Investigator — Baptist Health - Miami; Ajit Puri, MD, Principal Investigator — University of Massachusetts, Worcester; Thanh Nguyen, MD, Principal Investigator — Boston Medical Center
Locations (30):
- United States (29):
  - Banner Health, Mesa, Arizona
  - Mercy San Juan Medical Center, Carmichael, California
  - Christiana Care, Newark, Delaware
  - Baptist Jacksonville, Jacksonville, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Advocate Aurora Health, Chicago, Illinois
  - University of Kansas, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Tufts, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Saint Luke's, Kansas City, Missouri
  - Cooper Health System, Camden, New Jersey
  - Rutgers, Piscataway, New Jersey
  - Stony Brook University Hospital, Stony Brook, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health, Columbus, Ohio
  - Wright State University, Dayton, Ohio
  - Mercy Health St. Vincent, Toledo, Ohio
  - OHSU, Portland, Oregon
  - Geisinger Clinic, Danville, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - Fort Sanders Medical Center, Knoxville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - Valley Baptist, Harlingen, Texas
  - Medical City Plano, Plano, Texas
  - University of Utah, Salt Lake City, Utah
  - West Virginia University, Morgantown, West Virginia
- Auckland City Hospital, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nguyen TN, Dabus G, McGuinness B, Caldwell J, Priest R, Rai AT, Zaidat OO, Gross BA, Hanel R, Lee S, Hussain S, Shaikh H, Abdalkader M, Budzik R, Kilburg C, Woodward K, Colasurdo M, Liu J, Yoo AJ, Khandelwal P, Boo S, Vu P, Lin E, Almajali M, Singh J, Al-Bayati A, Lang MJ, Abraham M, Hassan AE, Pema P, Martin C, Grandhi R, Tonetti DA, Hixson HR, Aghaebrahim A, Sauvageau E, Ortega-Gutierrez S, Yavagal DR, Cheng-Ching E, Khalife J, Linfante I, Vulkanov V, Soomro J, Fifi JT, Maidan L, Copelan A, Schirmer CM, Bain M, Toth G, Jayaraman M, Novakovic-White R, Satti S, Villelli N, Jabbour P, Page M, McAllister DJ, Araujo Contreras R, Samaniego EA, Liebeskind DS, Hetts SW, Nogueira RG, English J, Puri AS. SUMMIT MAX: A Randomized Trial of the Super Large Bore HiPoint Reperfusion System Versus Vecta System for Aspiration Thrombectomy. Stroke. 2025 Aug;56(8):1980-1990. doi: 10.1161/STROKEAHA.125.051742. Epub 2025 May 21. PMID 40395106